CLINICAL TRIAL: NCT01941823
Title: Pilot Study: Effect of Carnitine Supplementation on Acylcarnitine Profile and Myocardial Function in Children and Young Adults Receiving Continuous Renal Replacement Therapy
Brief Title: Carnitine, Aclycarnitine, Myocardial Function, and CRRT
Status: Completed | Type: Observational
Sponsor: Asha Moudgil (Other)
Responsible Party: Sponsor-Investigator, Asha Moudgil, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: 00003555
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Acute Renal Failure
Keywords: acute renal failure; CRRT; continuous dialysis; carnitine; cardiac strain
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Carnitine CRRT, prospective: CRRT patients given carnitine in TPN as part of clinical protocol. Will evaluate total and free, carnitine and acylcarnitine profile as well as cardiac function by standard and speckle tracking echo weekly during CRRT.
- CRRT Control, retrospective: Retrospective control group, CRRT patients who did not receive carnitine supplementation during CRRT and had carnitine levels measured and echo performed during CRRT.
- ICU Control (non-CRRT), prospective: Critically ill ICU patients not receiving any exogenous carnitine, and not receiving CRRT, will have total and free carnitine and acylcarnitine profile measured weekly during CRRT.

SUMMARY:
Carnitine is essential for the transport of fatty acids into the mitochondria and energy production in different muscles, including the myocardium. It is also needed to protect myocyte cell membranes from oxidative damage by removing excess acyl carnitine groups. Patients receiving chronic intermittent hemodialysis (HD) are known to be at increased risk for carnitine deficiency as a result of its removal during the dialysis procedure, lack of endogenous synthesis by the kidney, and inadequate dietary intake. The carnitine status of children undergoing continuous renal replacement therapy (CRRT) has not been studied. Children undergoing CRRT in the intensive care unit (ICU) setting may be at increased risk for carnitine deficiency due to its continuous removal, lack of carnitine production by the kidney, and absence of carnitine intake (as majority of these children can not eat and there is no carnitine added to total parenteral nutrition (TPN). Carnitine deficiency may increase the risk of cardiac dysfunction in critically ill children. This is the first study to examine carnitine status in children undergoing CRRT. Standard echo as well as more sensitive speckle tracking echo will be used to evaluate the effect of carnitine deficiency on myocardial function.

DETAILED DESCRIPTION:
Study Design:The research design consists of a prospective study group that would be compared to two control groups (a prospective control groups and a retrospective control group). The study group will consist of critically ill children receiving CRRT and IV carnitine supplementation (added in the TPN). The prospective control group will consist of critically ill children not receiving CRRT or carnitine Retrospective control group will consist of critically ill children who received CRRT but did not receive carnitine supplementation. . Subjects for the prospective study and control groups will be recruited from the pediatric intensive care unit (PICU) and the cardiac intensive care unit (CICU) at Children's National. Informed consent will be obtained from participants enrolled in the prospective study and control groups. Data for the retrospective control group will be obtained from the medical record.

ELIGIBILITY:
Patients

CRRT Study Group (n=10) Inclusion Criteria

1. age 1-21 years
2. Receiving CRRT in the PICU or CICU
3. NPO or TPN-dependent Exclusion Criteria

1. Children on chronic dialysis 4. Children on carnitine supplementation for a metabolic disorder 5. Children on CRRT for less than 1 week

Prospective Control Group (n=10) Inclusion Criteria 1. age 1-21years 2. Receiving care in the PICU or CICU, but not requiring CRRT 3. NPO or TPN-dependent Exclusion Criteria

1. Children on chronic dialysis
2. Children on carnitine supplementation for a metabolic disorder

Retrospective CRRT Control Group (n=10) Inclusion Criteria

1. 1-21years of age
2. Received CRRT between 2011-2015
3. Had total and free carnitine level checked while on CRRT (2 values>1 week apart)
4. Had echocardiogram (2 studies >1 week apart) Exclusion Criteria

1. Receiving supplemental carnitine at time of carnitine level and/or echocardiogram 2. Congenital or acute heart disease 3. On ECMO

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young adults, age 1-21 years Critically ill, receiving care in intensive care unit
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2014-12; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Cardiac function of children receiving carnitine compared with controls during CRRT | 1-3 weeks
  Echocardiography parameters of children in the study group will be compared to those of the retrospective CRRT control group.

SECONDARY OUTCOMES:
Carnitine deficiency in children receiving CRRT | Baseline
  Total and free carnitine levels and acylcarnitine profile of the 3 study cohorts will be compared with published normal levels in children.

CONTACTS AND LOCATIONS:
Overall Officials: Asha Moudgil, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Cetner, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sgambat K, Moudgil A. Carnitine deficiency in children receiving continuous renal replacement therapy. Hemodial Int. 2016 Jan;20(1):63-7. doi: 10.1111/hdi.12341. Epub 2015 Aug 11. PMID 26265013